CLINICAL TRIAL: NCT05990517
Title: Evaluation of the Efficacy and Safety of Autologous Transplantation of Expanded Pancreatic Islet Cells (YD01-2022) in Patients With Diabetes Mellitus After Total Pancreatectomy
Brief Title: Autologous Transplantation of Expanded Pancreatic Islet Cells (YD01-2022) in Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YD01-2022
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes After Total Pancreatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YD01-2022 (Experimental)
  Interventions: Biological: YD01-2022

INTERVENTIONS:
Biological: YD01-2022 — Human islet cells were isolated and expanded in vitro to generate islets containing all types of pancreatic endocrine cells and possessing comparable function of human islets. These islet cells will be infused into the hepatic portal vein.

SUMMARY:
This study will evaluate the efficacy and safety of autologous transplantation of expanded pancreatic islet cells in patients with diabetes mellitus after total pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form and comply with the trial treatment plan and visit schedule.

2. Age ≥18 years and ≤60 years on the day of signing the informed consent form, regardless of gender.

3. Diagnosed with chronic pancreatitis and indication for total pancreatectomy. 4. Post-total pancreatectomy, experiencing elevated blood glucose levels and meeting the diagnostic criteria for diabetes (World Health Organization, 2019 edition).

5. Post-mixed meal stimulation, C-peptide level <0.3 ng/mL at 120 minutes. 6. Sexually active males who are not surgically sterilized or have partners of childbearing potential agree to use effective contraception during the entire trial period and for at least 6 months after the study ends; sexually active females of childbearing potential agree to use effective contraception during the entire study period and for at least 6 months after the study ends.

1. History of diabetes or preoperative diagnosis of hyperglycemia, meeting the diagnostic criteria for diabetes.
2. Previous pancreatic or islet transplantation.
3. Uncontrolled hypertension, such as systolic blood pressure (SBP) >160 mmHg and/or diastolic blood pressure (DBP) >100 mmHg despite stable dose (at least 4 weeks) of antihypertensive medication.
4. Known hemoglobin-related diseases, anemia (moderate to severe), or other known hemoglobinopathies that interfere with HbA1c measurement (such as sickle cell disease).
5. Impaired liver or kidney function at screening (reference range from the study center's laboratory): aspartate aminotransferase (AST) >3 times the upper limit of normal (ULN), alanine aminotransferase (ALT) >3 times ULN, total bilirubin level (TBL) >2 times ULN (excluding Gilbert's syndrome). Creatinine clearance rate <45 mL/min (calculated by the Cockcroft-Gault formula).
6. Significant albuminuria (urinary albumin excretion rate >300 mg/g) or history thereof.
7. Uncontrolled thyroid disease or adrenal insufficiency.
8. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA ≥104 copies or ≥2000 IU/mL (HBsAg positive with HBV DNA <2000 IU/mL (<104/mL) must receive antiviral treatment throughout the study; HBcAb positive with HBV DNA <2000 IU/mL (<104/mL) require regular monitoring of HBV DNA quantification throughout the study); Hepatitis C virus (HCV) antibody positive with peripheral blood HCV RNA ≥103 IU/mL; Human immunodeficiency virus (HIV) antibody positive; Active syphilis infection (cured cases may be included); Cytomegalovirus (CMV) DNA positive; Positive nucleic acid test for novel coronavirus (COVID-19).
9. Severe heart disease or a history of cardiovascular disease within 6 months before screening, including stroke, decompensated heart failure (NYHA class III or IV), myocardial infarction, unstable angina, or coronary artery bypass grafting.
10. Previous history of coagulation disorders or requiring long-term anticoagulant therapy (e.g., warfarin) (low-dose aspirin therapy is allowed) or patients with INR >1.5.
11. Substance abusers with a history of drug abuse/dependence or drug use within 1 year before screening.
12. Received live virus vaccines within the past 6 months or planned to receive live virus vaccines during the trial or within 1 month after treatment. Live vaccines include, but are not limited to, measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guérin, typhoid vaccine, COVID-19 vaccine, etc.
13. Previous history of pancreatic cancer, intraductal papillary mucinous neoplasm of the pancreas, end-stage lung disease, or liver cirrhosis.
14. Other abnormal laboratory test results deemed clinically significant by the investigator.
15. Patients with severe mental illness.
16. Participated in a drug or medical device clinical trial within the past 3 months and received investigational drugs or medical devices; or within 5 half-lives of another drug before screening (if the half-life exceeds 3 months).
17. Currently receiving long-term (continuous for ≥14 days) systemic pharmacological doses of glucocorticoids or other medications that may affect the participant's consciousness.
18. Treatment (local, intra-articular, intraocular, or inhalation preparations) for any other factors or diseases not mentioned above, deemed unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
C-peptide change | 12 months post-transplant
  Evaluation of the magnitude of C-peptide change after transplantation

SECONDARY OUTCOMES:
the proportion of subjects with HbA1c ≤7.0% and no severe hypoglycemic events | 52 weeks post-transplant
The proportion of subjects who are insulin-independent | 12 weeks and 52 weeks post-transplant
The percentage reduction in insulin requirement | 12 weeks and 52 weeks post-transplant
Glycemic control (MAGE) | 12 weeks and 52 weeks post-transplant
  Evaluation of the average amplitude of glycemic fluctuations (MAGE) in subjects
Evaluation of the severity of hypoglycemia using the Ryan Hypoglycemia Severity Score (HYPO) | baseline and 52 weeks post-transplant
Quality of life score | baseline and 52 weeks post-transplant
  Evaluation of the quality of life score in subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolic Diseases, Ruijin Hospital, Shanghai Jiao-Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided